CLINICAL TRIAL: NCT00949182
Title: Micro and Macro Arteriolar Blockade of Hepatocellular Carcinoma (HCC): Treatment With Sorafenib Before and After Hepatic Arterial Embolization (HAE) Therapy for Liver Cancer.
Brief Title: Sorafenib Tosylate Before and After Hepatic Arterial Chemoembolization With Doxorubicin Hydrochloride and Mitomycin C in Treating Patients With Localized Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Andrew de la Torre, M.D, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000649008; UMDNJ-20090859 (Other: WIRB); BAYER-IST000477 (Other Grant/Funding Number: Bayer Health Care Pharmaceuticals)
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Sorafenib; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib Tosylate, Doxorubicin, Mytomicin C (Experimental): Micro and Macro arteriolar blockade of hepatocellular carcinoma (HCC): Treatment with Sorafenib 400mg two weeks prior to embolization HACE which includes the use of agents such as Doxorubicin Hydrochloride and Mytomicin C, continuing same Sorafenib dose after the procedure (dose adjustment according to tolerance).
  Interventions: Drug: sorafenib tosylate, HACE : Doxorubicin Hydrochloride and Mitomycin C; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate, HACE : Doxorubicin Hydrochloride and Mitomycin C — After Sorafenib Tosylate has been administered the actual HACE procedure is performed using Doxorubicin Hydrochloride or Mitomycin C
  Other Names: Doxorubicin brand name Adriamycin.
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as doxorubicin hydrochloride and mitomycin C, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Chemoembolization kills tumor cells by carrying drugs directly into the tumor and blocking blood flow to the tumor. Giving sorafenib tosylate before and after chemoembolization may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving sorafenib tosylate before and after hepatic arterial chemoembolization with doxorubicin hydrochloride and mitomycin C works in treating patients with localized liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety and tolerability of sorafenib tosylate therapy when administered before and after doxorubicin hydrochloride-based hepatic arterial chemoembolization (HACE) as assessed by NCI CTCAE v3.0 in patients with localized unresectable hepatocellular carcinoma.

Secondary

* To determine if sorafenib tosylate decreases the number of HACE treatments required to achieve radiologic tumor kill.
* To assess improvement in progression-free survival.
* To assess changes in monthly AFP levels in patients with AFP-producing tumors.
* To measure VEGF levels.

OUTLINE: Patients receive oral sorafenib tosylate twice daily on days 1-14. Beginning ≥ 3 days later, patients undergo hepatic arterial chemoembolization (HACE)* with doxorubicin hydrochloride and mitomycin C. Beginning ≥ 3 days after the completion of HACE and/or once liver function returns to baseline, patients resume sorafenib tosylate twice daily for up to 6 months in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients may undergo more than one HACE treatment.

Blood samples are collected periodically for further laboratory analysis.

ELIGIBILITY:
Inclusion Criteria

* Age > 18 years old
* Confirmed HCC diagnosis by Biopsy or Radiologic parameters. Following NCCN guidelines for HACE, including subjects within the University of San Francisco transplant listing criteria.
* ECOG Performance Status 0 or 1
* Adequate bone marrow, liver and renal function as .assessed by the following:

  * Hemoglobin > 9.0 g/dl
  * Absolute neutrophil count (ANC) > 1,500/mm3
  * Platelet count > 75,000/mm3
  * Total bilirubin < 2 mg/dl
  * ALT and AST < 2.5 times the ULN ( < 5 x ULN for patients with liver involvement)
  * Creatinine < 1.5 times mg/dl
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* INR < 1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* BCLC Stage B (Intermediate)

  * multinodular asymptomatic tumors
  * without vascular invasion
  * without extrahepatic spread
* Child Pugh A through B7
* Male or female patients > 18 years of age
* Life expectancy of at least 12 weeks. Patients with unresectable, multinodular asymptomatic tumor (no vascular invasion or extrahepatic spread)
* Patients with histologically or cytologically documented HCC. Documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable
* Prior informed consent.
* At least one tumor lesion that meets both of the following criteria:

  * The lesion can be accurately measured in at least one dimension according to RECIST
  * The lesion has not been previously treated with local therapy (such as surgery, radiation therapy, RFA, PEI, or cryoablation)

Exclusion Criteria

* Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Known brain metastasis or CNS disease. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection
* Active clinically serious infection > CTCAE Grade 2 except hepatitis B or C.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.
* Use of any prior systemic chemotherapy or targeted agents.
* Diffuse HCC or presence of vascular invasion (including segmental portal obstruction), extrahepatic spread
* Advanced liver disease: unstable ascites or >Child-Pugh B7
* Porto-systemic shunt
* Any contraindication for an arterial procedure such as impaired clotting tests (platelet count < 50.000/mm3 or prothrombin activity < 50 percent), 1
* Renal failure
* Severe atheromatosis
* Any contraindication for systemic chemotherapy administration (serum bilirubin > 5mg/dL, leukocyte count < 3.000 cells/mm3)
* Any contraindication for sorafenib administration
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Pregnant or breast-feeding patients
* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated > 3 years prior to entry is permitted
* Patients receiving therapy for Hepatitis A, B or C
* Encephalopathy ≥ Grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by NCI CTCAE v3.0 | 06/2009 to 12/2010

SECONDARY OUTCOMES:
Number of hepatic arterial chemoembolization (HACE) treatments required to achieve objective complete response | 06/2009 to 12/2010
Progression-free survival and time to radiologic progression as assessed by CT scan | 06/2009 to 12/2010
Overall survival at 6, 12, and 24 months | 06/2009 to 12/2011
AFP and VEGF serum levels as assessed at baseline, prior to each HACE treatment, and then every 3 months thereafter | 06/2009 to 12/2011

CONTACTS AND LOCATIONS:
Overall Officials: Andrew N. de la Torre, MD, Principal Investigator — Rutgers University Hospital / St Joseph Medical Center
Locations (1):
- Rutgers University Hospital, Newark, New Jersey, United States